CLINICAL TRIAL: NCT04828603
Title: Understanding Allergies
Brief Title: Understanding Allergies and Sensitizations in Healthy and Allergic Individuals
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Crown Fundation (Unknown); Sunshine Foundation (Unknown); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Human Genome Research Institute (NHGRI) (NIH); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, Associate Professor & Director, Clinical Translational Research Unit, Stanford University
Other Study IDs: 8629; 1R01AI165866-01 (NIH); 1DP2HG012480-01 (NIH)
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples; additional samples could include sputum, urine sample, stool sample, oral and nasal samples, skin samples, gastrointestinal samples, and surgical tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to strengthen our ability to accurately diagnose allergies and understand cellular, humoral, genetic components and physiological changes in allergic disease

ELIGIBILITY:
Inclusion Criteria:

* Any individual with possible allergy

Exclusion Criteria:

* Patients with special risks attendant to venipuncture will be excluded

Ages: 1 Week to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients ages 1 week through 90 years who have or are suspected of having allergic sensitivities will be invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2007-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Skin testing to evaluate food allergen responses | 1 year
  Standardized skin testing performed to detect sensitivity to allergens of interest

CONTACTS AND LOCATIONS:
Overall Officials: R. Sharon Chinthrajah, MD, Principal Investigator — Stanford University
Locations (1):
- Sean N. Parker Center for Allergy and Asthma Research, Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No